CLINICAL TRIAL: NCT05994066
Title: Effect of Sleep Quality,Physical and Mental Fatigue on Mechanical Neck Pain
Brief Title: Sleep Disturbance,Physical and Mental Fatigue on Mechanical Neck Pain
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Zeinab Abd el fattah Ali, assistant professor, Cairo University
Other Study IDs: Sleep disturbance,physical and
Record Dates: First submitted 2023-08-08; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Mechanical Neck Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Demographic data of the individuals were recorded. All participants completed NDI, Chalder Fatigue Scale (CFS) and Pittsburgh Sleep Quality Index (PSQI). — Demographic data of the individuals were recorded. All participants completed NDI, Chalder Fatigue Scale (CFS) and Pittsburgh Sleep Quality Index (PSQI).

SUMMARY:
Mechanical neck pain is a prevalent problem in community and it can lead to disability.

In current community, increasing of life stress on individual may lead to sleep disorders, mental and physical fatigue.

Objectives of study is to investigate the effect of sleep quality, mental and physical fatigue on mechanical neck pain.

Methods and Materials Two hundred thirty individuals were having mechanical neck pain . Neck disability index, chalder fatigue scale and Pittsburg sleep quality index were applied on all individuals participating in the study , NDI was used to determine the pain and functional disability of the participants , PSQI was used to assess the sleep quality, lastly the CFS was used to determine

DETAILED DESCRIPTION:
Our study considered as an observational cross - sectional study.

Sample size :

Individual's ;230 patient with mechanical neck pain will participate in the study The inclusion criteria were age between 18 -60 years , who do have neck disability index score more than (4) points, they have being included in our study. The exclusion criteria were people who are having any cervical injury( fracture,whiplash injury) cervical disc , neurological disease, past surgery in neck region. Also we excluded who has been scored with 4 points or less in NDI . The study will be in the out clinic of orthopedic in faculty of physical therapy , cairo university

Material tool :

We used three index , NECK DISABILITY INDEX [NDI] , CHALDER FATIGUE SCALE [CFS] , PITTSBURGH SLEEP QUALITY SCALE [PSQI]. -NDI : neck disability index is consists of 10 questions including = pain severity,ability of personal care ,lifting weight, job capability, headaches intense , concentration, quality of sleeping and driving and recreation activities. The total score ranges between 0- 50 points . Zero to 4 points mean( NO DISABILITY), 5 to 14 points means (LIGHT DISABILITY ) , 15 to 24 points means ( MODERATE DISABILITY ), 25 to 34 points means (SEVERE DISABILITY) 35 to 50 points means (COMPLETE DISABILITY).

- CFS : The CFS is consisting of 11 questions including a seven item physical fatigue subdimension and a four item mental fatigue sub-dimension.The physical fatigue subdimension score ranges from 0 to 21, the mental fatigue sub-dimension score from 0 to12 The total fatigue score is from 0-33. High scores indicates a greater fatigue level.

- PSQI : The scale is consisting of 24 items,19 items are filled by the individuals,while 5 are filled by the bedmate*if they have one*. 18 of 19 items that filled by the individual himself

\herself are scored and used to asses sleep quality,while the remaining 6 items are used to have clinical inflammation. It has 7 components:

1. subjective sleep quality
2. sleep latency
3. sleep duration
4. habitual sleep efficiency
5. sleep disturbances
6. use of sleeping pills
7. day time dysfunction . The total PUKIN score is obtained by summing the score of the components. The total of each item is 0-3 while the total score of PUKI is ranging between 0-21 . High score indicates poor sleep quality. A total score of 5 or less is indicating good sleep quality, while scores above 5 indicates poor sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were age between 18 -60 years , who do have neck disability index score more than (4) points, they have being included in our study.

Exclusion Criteria:

* The exclusion criteria were people who are having any cervical injury( fracture,whiplash injury) cervical disc , neurological disease, past surgery in neck region. Also we excluded who has been scored with 4 points or less in NDI

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Our study considered as an observational cross - sectional study. 230 patients will participate in the stuudy The inclusion criteria will be age between 18 -60 years , who do have neck disability index score more than (4) points, they have being included in our study. The exclusion criteria were people who are having any cervical injury( fracture,whiplash injury) cervical disc , neurological disease, past surgery in neck region. Also we excluded who has been scored with 4 points or less in NDI . The study was on online survey we used what'sup app and telegram app
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2023-08-30 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Arabic version of NDIto determine the pain experience and functional disability of the participants. | 1 month
  NDI consists of 10 questions concern of the pain severity, ability for personal care, lifting weight, job capability headache intensity, concentration, quality of sleeping and driving and recreation activities. Total score ranges between 0 to 50 points. Zero to four points mean "no disability", 5 to 14 points mean "light disability", 15 to 24 points mean "moderate disability", 25 to 34 points mean "severe disability", and 35 to 50 points mean "complete disability" (15).
Pittsburgh Sleep Quality Index (PSQI) | 1 month
  In this scale consisting of 24 items, 19 items are filled in by the individual, while five items are filled in by the person's bedmate. Eighteen of the 19 items that need to be answered by the individual are scored and used to assess sleep quality, while the remaining six items are used to have clinical information. It has seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping pills, and daytime dysfunction. The total PUKI score is obtained by summing the scores of the components. The total score of each component varies between zero to three and the total score of PUKI ranges from 0 to 21. High scores indicate poor sleep quality. A total score of five or less indicates good sleep quality, while scores above 5 indicate poor sleep quality (16).
Chalder Fatigue Scale (CFS) | 1 month
  CFS consists of 11 questions including a 7-item physical fatigue sub-dimension and a 4-item mental fatigue sub-dimension (19). 4-point Likert scale was used. The scoring of each item varies between zero to three points. The physical fatigue sub-dimension score ranges from 0 to 21, the mental fatigue sub-dimension score ranges from 0 to 12, and the total fatigue score ranges from 0 to 33. High scores indicate a greater fatigue level (18). The arabic version of the questionnaire was used in the study (19).

CONTACTS AND LOCATIONS:
Overall Officials: zeinab Ali, phd, Principal Investigator — Cairo University

REFERENCES:
- [Background] Bonvanie IJ, Oldehinkel AJ, Rosmalen JGM, Janssens KAM. Sleep problems and pain: a longitudinal cohort study in emerging adults. Pain. 2016 Apr;157(4):957-963. doi: 10.1097/j.pain.0000000000000466. PMID 26683236
- [Background] Bjornsdottir SV, Jonsson SH, Valdimarsdottir UA. Mental health indicators and quality of life among individuals with musculoskeletal chronic pain: a nationwide study in Iceland. Scand J Rheumatol. 2014;43(5):419-23. doi: 10.3109/03009742.2014.881549. Epub 2014 May 12. PMID 24814312